CLINICAL TRIAL: NCT01961687
Title: A Prospective, Multi-Center Study of Phasix™ Mesh for Ventral or Incisional Hernia Repair.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DVL-HE-011
Record Dates: First submitted 2013-10-10; First posted 2013-10-11 (Estimated); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Ventral Hernia; Incisional Hernia
MeSH Terms: conditions — Hernia, Ventral; Incisional Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Resorbable Mesh (Other): Phasix Mesh
  Interventions: Device: Resorbable Mesh

INTERVENTIONS:
Device: Resorbable Mesh — Phasix Mesh

SUMMARY:
Single-arm study of Phasix Mesh in High Risk patients looking at SSI and recurrence rates.

DETAILED DESCRIPTION:
The objective of this study is to collect additional data on safety, performance and effectiveness of Phasix™ Mesh in subjects requiring primary ventral, incisional or first-recurrent (protocol version 1.4)/multiply-recurrent (protocol version 2.0) hernia repair in subjects at high risk for complications. Subjects at high risk are defined as having 1 or more of the following co-morbidity conditions: body mass index (BMI) between 30-40 kg/m2, inclusive, active smokers, chronic obstructive pulmonary disease (COPD), diabetes, immunosuppression, coronary artery disease, chronic corticosteroid use, low pre-operative serum albumin, advanced age, or renal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

Subjects must have met all of the criteria listed below to be enrolled in the study:

1. Subject must have been 18 years of age or older 2. Subject or subject's legally authorized representative must have given written informed consent 3. Subject must have been diagnosed with primary ventral, incisional hernia or first time recurrent ventral or incisional hernia (protocol version 1.4) 3. Subject must be diagnosed with primary ventral, incisional hernia or multiply-recurrent (not to exceed 3 recurrences) ventral or incisional hernia (protocol version 2.0) 4. Subject must have had a hernia greater than 10 cm2 and ≤350 cm2 5. Subject must have been willing to undergo initial ventral, incisional or first recurrent incisional hernia repair using retro-rectus or onlay placement (using absorbable suture) with or without Component Separation Technique (CST) (protocol version 1.4) 5. Subject must be willing to undergo initial ventral, incisional or multiply-recurrent incisional hernia repair using retro-rectus or onlay placement (using absorbable suture) with or without Component Separation Technique (CST) (protocol version 2.0) 6. Subject met the criteria for a Class I wound as defined by the CDC (Appendix 4 of the protocol) 7. Subjects must have had 1 or more of the following pre-study conditions:

1. Body Mass Index (BMI) between 30-40 kg/m2, inclusive
2. Active smokers (if attempts to quit smoking within two weeks of surgery have failed and the patient was still an active smoker at the time of surgery)
3. COPD presence on patient self-report
4. Diabetes mellitus
5. Immunosuppression
6. Coronary Artery Disease
7. Chronic corticosteroid use: greater than 6 months systemic use
8. Serum albumin less than 3.4 g/dL
9. Advanced age: 75 years or older
10. Renal insufficiency, defined as serum creatinine concentration ≥2.5 mg/dL

Exclusion Criteria:

Subjects were excluded from study enrollment if any of the following criteria were met:

1. Subject's hernia had recurred more than once (protocol version 1.4)

1. Subject has had 4 or more previous hernia repairs (of the index hernia) (protocol version 2.0)
2. The subject had peritonitis
3. The subject was on or suspected to be placed on chemotherapy medications during any part of the study
4. The subject's Body Mass Index (BMI) was greater than 40 kg/m2
5. The subject had cirrhosis of the liver and/or ascites
6. Subject was American Society of Anesthesiology Class 4 or 5
7. Subject was known to be infected with human immunodeficiency virus (HIV)
8. Subject had a life expectancy of less than 2 years at the time of enrollment
9. Subject had any condition that, in the opinion of the Investigator, precluded the use of the study device, precluded the subject from completing the follow-up requirements
10. Subject's hernia repair utilized intraabdominal mesh placement
11. Subject had a surgical wound classified as Class II (Clean-Contaminated), Class III (Contaminated) or Class IV (Dirty-Contaminated) as defined by the CDC (Appendix 4 of the protocol)
12. Subject had an active or latent systemic infection
13. Subject required surgical bridge repair as the sole repair
14. Subject was pregnant or had plans to become pregnant during the study period or was breastfeeding
15. Subject had enrolled in another clinical study within the last 30 days
16. Subject was part of the site personnel directly involved with this study
17. Subject had a known allergy to the test device or component materials (patients with known allergies to tetracycline hydrochloride or kanamycin sulfate were avoided).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Roth, MD, Principal Investigator — University of Kentucky
Locations (16):
- United States (16):
  - University of California, San Diego, San Diego, California
  - Florida Hospital/Celebration Health, Celebration, Florida
  - NorthShore University HealthSystem, Evanston, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - Methodist Health System, Omaha, Nebraska
  - Southeast Area Health and Education Center, Wilmington, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Univerity of Tennessee Health Science Center, Germantown, Tennessee
  - University of Tennessee Health Sciences Center, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Wisconsin System, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roth JS, Anthone GJ, Selzer DJ, Poulose BK, Pierce RA, Bittner JG, Hope WW, Dunn RM, Martindale RG, Goldblatt MI, Earle DB, Romanelli JR, Mancini GJ, Greenberg JA, Linn JG, Parra-Davila E, Sandler BJ, Deeken CR, Badhwar A, Salluzzo JL, Voeller GR. Long-Term, Prospective, Multicenter Study of Poly-4-Hydroxybutyrate Mesh (Phasix Mesh) for Hernia Repair in Cohort at Risk for Complication: 60-Month Follow-Up. J Am Coll Surg. 2022 Dec 1;235(6):894-904. doi: 10.1097/XCS.0000000000000363. Epub 2022 Nov 15. PMID 36102523

RESULTS

PARTICIPANT FLOW:
Groups:
- Phasix Mesh Group: Patients requiring primary ventral, incisional, or recurrent hernia repair at high risk for complications. Subjects defined to be at high risk must have one or more of the following conditions pre-study: body mass index (BMI) between 30-40 kg/m2 inclusive, be an active smoker, have chronic obstructive pulmonary disease (COPD), diabetes mellitus, immunosuppression, coronary artery disease, chronic corticosteroid use (>6 months systemic use), serum albumin ≤3.4 g/dL, age over 75 years, or renal insufficiency (defined as serum creatinine concentration ≥2.5 mg/dL).
Period: Overall Study
Arm/Group | Phasix Mesh Group
Started | 121
Completed | 60
Not Completed | 61
Not completed — Lost to Follow-up | 19
Not completed — Re-operation | 17
Not completed — Death | 7
Not completed — Withdrawal by Subject | 6
Not completed — Adverse Event | 6
Not completed — Moved to area without study site | 2
Not completed — Sponsor decision | 2
Not completed — Physician Decision | 1
Not completed — Unable to meet follow-up requirements | 1

BASELINE CHARACTERISTICS:
Groups:
- Phasix Mesh: Subjects requiring primary ventral, incisional, or recurrent hernia repair at high risk for complications. Subjects defined to be at high risk must have one or more of the following conditions pre-study: body mass index (BMI) between 30-40 kg/m2 inclusive, be an active smoker, have chronic obstructive pulmonary disease (COPD), diabetes mellitus, immunosuppression, coronary artery disease, chronic corticosteroid use (>6 months systemic use), serum albumin ≤3.4 g/dL, age over 75 years, or renal insufficiency (defined as serum creatinine concentration ≥2.5 mg/dL).
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 94
  >=65 years | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 113
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 116
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 121
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.24 (4.52)

OUTCOME MEASURES:

1. Primary Outcome: Hernia Recurrence Rate
Description: Hernia recurrence rates will be assessed by physical examination at each study visit through 60 months. A recurrent hernia will be defined as any hernia identified or confirmed by the investigator, during any study follow-up visit, in approximately the same position as the hernia repaired in the study procedure. Potential hernias identified via incidental magnetic resonance imaging (MRI) or computed tomography (CT) scan will be evaluated by the operating surgeon for clinical significance and confirmation of hernia recurrence.
Time Frame: 60 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 121
Participants | 20

2. Primary Outcome: Surgical Site Infections
Description: Infections at the surgical site will be assessed by physical examination at each study visit through 60 months. If an infection is suspected, a routine culture, obtained via each site's standard protocol, should be obtained to determine cell count and type (i.e. yeast, gram positive or gram negative bacteria, or other). If genus and species of the culture are identified as part of the routine practice at the site, that information should be recorded. Classification will follow the CDC guidelines for superficial and deep surgical site infections
Time Frame: 60 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 121
Participants | 11

3. Secondary Outcome: Pain Visual Analog Scale
Description: Mean change in self-reported pain measured on a Visual Analog Scale between Baseline and 60-month follow up. Scores are measured on a scale from 0.0 to 10.0 centimeters and marked on a line by the subject; lower values correspond with low pain perception. The outcome measure is presented as the mean of the absolute difference between the pain perception at Baseline and the pain perception at 60-month follow up. A negative score means a decrease in pain perception.
Time Frame: 60 Months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 121
cm | -3.16 (3.35)

4. Secondary Outcome: Device Related Adverse Events
Description: Incidence of device related adverse events: number of subjects with one or more possibly or definitely device related adverse events. The term "incidence" is an error and is reported here as the rate of device related adverse events.
Time Frame: 60 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 121
Participants | 19

5. Secondary Outcome: Rate of Re-operation Due to the Index Hernia Repair
Description: Rate of re-operation due to the index hernia repair; the proportion of subjects with post-procedure re-operation due do the index hernia repair.
Time Frame: 60 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 121
Participants | 18

6. Secondary Outcome: Carolinas Comfort Scale® (CCS)
Description: Each scale score (sensation of mesh, pain or movement limitations) ranges from 0-5 and is a summation of scores across the domains. Therefore, the Total CCS Score ranges from 0-115 and is the average of the 3 scale scores. Low scores represent fewer symptoms or difficulties.
  Absolute values of the Total CCS Score at 1-Month follow-up, at 3-Month follow-up, at 6-Month follow-up, 12-Month follow-up, 18-Month follow up, at 24-Month follow-up, 36-Month follow-up, 48-Month follow-up, and 60-Month follow-up are reported.
  The absolute value at Baseline, or a change in self-reported quality of life measured by Carolinas Comfort Scale® cannot be reported, as subjects had incorrectly answered the questions on Sensation of Mesh at Baseline where no Phasix Mesh was yet implanted, thereby creating a bias in the results.
Time Frame: 60 Months
Population: The number of participants noted at each time point differ from the overall number (121) due to only having the eligible questionnaires being analyzed. The number of eligible questionnaires range from 52 to 111.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 121
Score on a scale
  Total CCS Score at 1 Month: number analyzed (Participants) | 111
  Total CCS Score at 1 Month | 31.2 (23.3)
  Total CCS Score at 3 Month: number analyzed (Participants) | 111
  Total CCS Score at 3 Month | 18.5 (20.9)
  Total CCS Score at 6 Month: number analyzed (Participants) | 109
  Total CCS Score at 6 Month | 14.1 (20.7)
  Total CCS Score at 12 Month: number analyzed (Participants) | 100
  Total CCS Score at 12 Month | 11.6 (21.1)
  Total CCS Score at 18 Month: number analyzed (Participants) | 93
  Total CCS Score at 18 Month | 8.4 (16.6)
  Total CCS Score at 24 Month: number analyzed (Participants) | 89
  Total CCS Score at 24 Month | 10.5 (20.7)
  Total CCS Score at 36 Month: number analyzed (Participants) | 80
  Total CCS Score at 36 Month | 9.8 (21.4)
  Total CCS Score at 48 Month: number analyzed (Participants) | 55
  Total CCS Score at 48 Month | 9.8 (21.4)
  Total CCS Score at 60 Month: number analyzed (Participants) | 52
  Total CCS Score at 60 Month | 4.9 (14.2)

7. Secondary Outcome: SF-12 Questionnaire
Description: The Short Form (SF)-12 version 2 (v2) is a multi-purpose, twelve item health survey that measures seven domains of health: general health, physical functioning, role limitations due to physical health (role-physical), role limitations due to emotional problems (role-emotional), bodily pain, vitality and mental health and social functioning. The SF-12v2 yields scale scores for each of these seven health domains, and two summary measures of physical and mental health: the physical component summary (PCS) and mental component summary (MCS). The scores range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: 60 Months
Measure: Mean (Standard Deviation); unit: Absolute Change from Baseline
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 121
Absolute Change from Baseline
  PCS - Month 1 | -2.700 (9.999)
  PCS - Month 3 | 5.374 (8.951)
  PCS - Month 6 | 6.943 (9.352)
  PCS - Month 12 | 6.868 (10.986)
  PCS - Month 18 | 7.589 (11.416)
  PCS - Month 24 | 6.206 (10.442)
  PCS - Month 36 | 7.101 (9.652)
  PCS - Month 48 | 7.206 (12.045)
  PCS - Month 60 | 7.374 (9.997)
  MCS - Month 1 | 0.546 (10.304)
  MCS - Month 3 | 3.287 (9.822)
  MCS - Month 6 | 3.311 (9.911)
  MCS - Month 12 | 2.124 (9.648)
  MCS - Month 18 | 2.015 (11.183)
  MCS - Month 24 | 2.769 (9.841)
  MCS - Month 36 | -0.239 (11.142)
  MCS - Month 48 | 2.393 (10.240)
  MCS - Month 60 | 3.248 (10.782)

8. Secondary Outcome: Surgical Procedure Time as Measured From Incision to Closure
Description: Surgical procedure time as measured from incision to closure (skin to skin)
Time Frame: 1 day
Measure: Mean (Full Range); unit: Minutes
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 121
Minutes | 168 [34 to 441]

9. Secondary Outcome: Length of Hospital Stay
Description: Time in days from hospital admission to discharge
Time Frame: 35 days
Measure: Median (Full Range); unit: Days
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 121
Days | 4 [1 to 35]

ADVERSE EVENTS:
Time Frame: 60 Months
Description: In this study, an Adverse Event (AE) is defined as any undesirable clinical event occurring in the abdominal space including the lower abdominal, inguinal and pubic regions (including the skin), as well as any other undesirable clinical events judged to be related to the study device or surgical procedure regardless of anatomical region. The definition of Serious AE does not deviate.
  Monitors have actively reviewed the subjects' medical records for Adverse Events during monitor visits.
Arm/Group | Phasix Mesh
All-Cause Mortality (participants affected / at risk) | 7/121
Serious Adverse Events (participants affected / at risk) | 49/121
Other Adverse Events (participants affected / at risk) | 104/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phasix Mesh (N=121)
Cardiac Arrest (Cardiac disorders) | 2 (2)
Cardiac Failure Acute (Cardiac disorders) | 1 (1)
Cardio-respiratory Arrest (Cardiac disorders) | 1 (1)
Right Ventricular Failure (Cardiac disorders) | 1 (1)
Abdominal Adhesions (Gastrointestinal disorders) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Abdominal Wall Disorder (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Colonic Pseudo-obstruction (Gastrointestinal disorders) | 1 (1)
Food Poisoning (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 (2)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1)
Hiatus Hernia (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 2 (2)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Peptic Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 5 (8)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 2 (2)
Generalized Oedema (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cholecystitis Chronic (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 1 (1)
Abdominal Abscess (Infections and infestations) | 1 (2)
Clostidium Deficile Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Post-operative Wound Infection (Infections and infestations) | 5 (5)
Sepsis (Infections and infestations) | 2 (2)
Septic Shock (Infections and infestations) | 2 (2)
Abdominal Wound Dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Cardiac Valve Replacement Complication (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1)
Incision Site Erythema (Injury, poisoning and procedural complications) | 1 (1)
Incision Site Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Incisional Hernia (Injury, poisoning and procedural complications) | 12 (12)
Incisional Hernia, Obstructive (Injury, poisoning and procedural complications) | 1 (1)
Joint Dislocation (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 2 (2)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 2 (2)
Skin Flap Necrosis (Injury, poisoning and procedural complications) | 1 (1)
Ureteric Injury (Injury, poisoning and procedural complications) | 1 (1)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pseudomyxoma Peritonei (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Embolic Cerebral Infarction (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (3)
Hemiparesis (Nervous system disorders) | 1 (1)
Hemiplegia (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Serotonin Syndrome (Nervous system disorders) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 2 (2)
Adnexa Uteri Cyst (Reproductive system and breast disorders) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Restrictive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin Necrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 2 (3)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Intra-abdominal Haematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phasix Mesh (N=121)
Abdominal Pain (Gastrointestinal disorders) | 26 (30)
Constipation (Gastrointestinal disorders) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 7 (7)
Ileus (Gastrointestinal disorders) | 8 (8)
Nausea (Gastrointestinal disorders) | 14 (15)
Vomiting (Gastrointestinal disorders) | 7 (8)
Postoperative Wound Infection (Infections and infestations) | 6 (6)
Abdominal Wound Dehiscence (Injury, poisoning and procedural complications) | 19 (20)
Incisional Hernia (Injury, poisoning and procedural complications) | 11 (12)
Procedural Pain (Injury, poisoning and procedural complications) | 14 (14)
Seroma (Injury, poisoning and procedural complications) | 11 (13)
Urinary Retention (Renal and urinary disorders) | 6 (7)

LIMITATIONS AND CAVEATS:
The study was designed as a single arm observational trial without pre-defined statistical hypotheses (theories) to test; therefore, data can only be described and no treatment or conclusions can be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT01961687/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT01961687/SAP_001.pdf